CLINICAL TRIAL: NCT04033861
Title: Prospective Observational Clinical Study：The Impact of Early rhBNP on Myocardial Remodeling and Reperfusion in Patients With ST-segment Elevation Myocardial Infarction After Percutaneous Coronary Intervention
Brief Title: Early rhBNP on Myocardial Remodeling and Reperfusion in Patients With STEMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai 6th People's Hospital (Other); Shanghai Minhang Central Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Suqian First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rhBNP-myocardium
Record Dates: First submitted 2019-01-24; First posted 2019-07-26 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2022-12

CONDITIONS: ST Segment Elevated Myocardial Infarction
Keywords: ST Segment Elevated Myocardial Infarction; rhBNP; cardiac magnetic resonance; Microvascular disease; ventricular remodeling
MeSH Terms: conditions — Ventricular Remodeling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhBNP (Experimental): rhBNP intra-coronary injection 1.5 ug/kg loading dose, with intravenous injection 0.0075-0.01 ug/kg/min persistent for 72 hour.
  Interventions: Drug: rhBNP
- Control (Placebo Comparator): saline intra-coronary injection 0.15ml/kg loading dose, with same intravenous injection speed for 72 hour after randomization.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: rhBNP — rhBNP intra-coronary injection 1.5 ug/kg loading dose, with intravenous injection 0.0075-0.01 ug/kg/min persistent for 72 hour.
  Arms: rhBNP
Drug: Control — saline intra-coronary injection 0.15ml/kg loading dose, with same intravenous injection speed for 72 hour.
  Arms: Control

SUMMARY:
The study intends to evaluate the efficacy of early rhBNP on myocardial remodeling and reperfusion in patients with ST-segment elevation myocardial infarction after percutaneous coronary intervention

DETAILED DESCRIPTION:
As prospectively observational study，it brings anterior acute myocardial infarct patients from 2018 JAN. to 2019 JAN, whose predefined time between symptom onset and percutaneous is not more than 12 hours. The door-to-balloon time, present to balloon time and first medical contact-to-balloon time will be documented. ECG in FMC and 90min after PCI also will be record. Patients assigned to the rhBNP group will receive intravenous rhBNP before PCI，and the variety of heart rate and blood pressure will be record. Routinely evaluation of corrected TIMI frame counting（CTFC）, TIMI myocardial perfusion frame counting and TIMI myocardial perfusion grade(TMPG).Blood tests including BNP, CK-MB and CRP are measured at admission and6, 12, 24, 48 hours after PCI. Both Cardiovascular magnetic imaging and echocardiography will be applied in Day 30 and 12 months. The composite endpoint is incidence of all-cause mortality, reinfarct, stroke and target vessel revascularization at hospitalization and follow-up. Principally patients are prevented from any drug affecting microcirculation (GPIIb/IIa receptor agonist, vascular dilation drug, etc.), otherwise it is necessary, which should be documented.

ELIGIBILITY:
Patients are eligible for enrollment if they are suspected as anterior myocardial infarct (anterior myocardial infarct is defined as persistent chest pain for 30 mins at least, with ST-segment elevation of at least 0.2 mV in two or more contiguous precordial leads) within 12 hours after onsets of symptom, and no contraindication for rhBNP. The coronary angiography (CAG) proves left anterior descending (LAD) as culprit vessel, which was totally or nearly occlusion with TIMI 0-1 grade and resulted in TIMI 3 grade after PCI.

Exclusive criteria:

1. Killips grade III-IV.
2. unstable hemodynamic; with A-V block or atrial fibrillation;
3. Contraindication of magnetic resonance, such as history of metal, ICD or paceman implant;
4. history of myocardial infarct;
5. pregnancy or breeding;
6. combined with other serious diseases: severe renal dysfunction (creatinine clearance<30ml/min;), liver failure, neutropenia, thrombocytopenia, acute pancreatitis；
7. life expectancy≤12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Compound endpoints of epicardium and endocardium perfusion | 90min after infarct related artery revascularization
  Both the TIMI and TMPG score reach 3 immediately after PCI, besides ST resolution≥70% at 90min after PCI.

SECONDARY OUTCOMES:
ST-segment Resolution | 90 mins after PCI
  Resolution of the initial sum of ST-segment elevation ≥ 70%
Wall motion score index (WMSI) and LVEF by echocardiography | Day 1, 3, 7, 30 and 12 month after PCI
  Echocardiographic index includes WMSI and LVEF
TIMI Flow Grade (TFG) | One mins after PCI
  TIMI Flow Grade (TFG)assesses flow in the epicardial arteries
TIMI Frame Count (CTFC) | One mins after PCI
  CTFC is a continuous measurement assessing flow in the epicardial arteries.
TIMI Myocardial Perfusion Grade (TMPG) | One mins after PCI
  TMPG is an angiographic measure of myocardial perfusion
TIMI Myocardial Perfusion Frame Count (TMPFC) | One mins after PCI
  TMPFC is a novel method to standardize and quantify myocardial perfusion by timing the filling and washout of contrast in the myocardium using cine-angiographic frame-counting. Briefly, the first frame of TMPFC was defined as the frame that clearly demonstrated the first appearance of myocardial blush beyond the IRA (F1). The last frame of TMPFC was then defined as the frame where contrast or myocardial blush disappeared (F2). TMPFC is F2-F1 frame counts at a filming rate of 15 frames/sec, or (F2-F1)×2 frame counts at the corrected filming rate of 30 frames/sec
CMR imaging | Day 1, 3, 7, 30 and 12 month after PCI
  CMR imaging will be collected using a 3.0-Tesla-scanner (Achieva, Philips Healthcare, The Netherlands) under electrocardiogram-triggered gating in School Shanghai Jiaotong University school of medicine RenJi hospital.

OTHER OUTCOMES:
hemodynamic adverse related to rhBNP | 72 hour since rhBNP administration
  low perfusion sign, and Noninvasive systolic blood pressure is below 90mmHg with or without diastolic blood pressure below 60mmHg, Excluding other reason.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD,PhD, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong Univers
Locations (1):
- Ren Ji Hospital Afflited to School of Medicine, Shanghai Jiao Tong University, Shanghai, China

REFERENCES:
- [Background] Ding S, Pu J, Qiao ZQ, Shan P, Song W, Du Y, Shen JY, Jin SX, Sun Y, Shen L, Lim YL, He B. TIMI myocardial perfusion frame count: a new method to assess myocardial perfusion and its predictive value for short-term prognosis. Catheter Cardiovasc Interv. 2010 Apr 1;75(5):722-32. doi: 10.1002/ccd.22298. PMID 19960517
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Gibson CM, Cannon CP, Murphy SA, Ryan KA, Mesley R, Marble SJ, McCabe CH, Van De Werf F, Braunwald E. Relationship of TIMI myocardial perfusion grade to mortality after administration of thrombolytic drugs. Circulation. 2000 Jan 18;101(2):125-30. doi: 10.1161/01.cir.101.2.125. PMID 10637197
- [Background] van 't Hof AW, Liem A, Suryapranata H, Hoorntje JC, de Boer MJ, Zijlstra F. Angiographic assessment of myocardial reperfusion in patients treated with primary angioplasty for acute myocardial infarction: myocardial blush grade. Zwolle Myocardial Infarction Study Group. Circulation. 1998 Jun 16;97(23):2302-6. doi: 10.1161/01.cir.97.23.2302. PMID 9639373
- [Background] Chinese Society of Cardiology of Chinese Medical Association; Editorial Board of Chinese Journal of Cardiology. [Guideline of non-ST segment elevation acute coronary syndrome]. Zhonghua Xin Xue Guan Bing Za Zhi. 2012 May;40(5):353-67. No abstract available. Chinese. PMID 22883082
- [Background] Kidambi A, Mather AN, Motwani M, Swoboda P, Uddin A, Greenwood JP, Plein S. The effect of microvascular obstruction and intramyocardial hemorrhage on contractile recovery in reperfused myocardial infarction: insights from cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2013 Jun 27;15(1):58. doi: 10.1186/1532-429X-15-58. PMID 23806080
- [Background] Roe MT, Ohman EM, Maas AC, Christenson RH, Mahaffey KW, Granger CB, Harrington RA, Califf RM, Krucoff MW. Shifting the open-artery hypothesis downstream: the quest for optimal reperfusion. J Am Coll Cardiol. 2001 Jan;37(1):9-18. doi: 10.1016/s0735-1097(00)01101-3. PMID 11153779
- [Background] Pu J, Shan P, Ding S, Qiao Z, Jiang L, Song W, Du Y, Shen J, Shen L, Jin S, He B. Gender differences in epicardial and tissue-level reperfusion in patients undergoing primary angioplasty for acute myocardial infarction. Atherosclerosis. 2011 Mar;215(1):203-8. doi: 10.1016/j.atherosclerosis.2010.11.019. Epub 2010 Nov 26. PMID 21176835
- [Background] Pu J, Ding S, Shan P, Qiao Z, Song W, Du Y, Shen J, Jin S, He B. Comparison of epicardial and myocardial perfusions after primary coronary angioplasty for ST-elevation myocardial infarction in patients under and over 75 years of age. Aging Clin Exp Res. 2010 Aug;22(4):295-302. doi: 10.1007/BF03337726. Epub 2009 Dec 1. PMID 20009495
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Shen LH, Wan F, Shen L, Ding S, Gong XR, Qiao ZQ, Du YP, Song W, Shen JY, Jin SX, Pu J, Yao TB, Jiang LS, Li WZ, Zhou GW, Liu SW, Han YL, He B. Pharmacoinvasive therapy for ST elevation myocardial infarction in China: a pilot study. J Thromb Thrombolysis. 2012 Jan;33(1):101-8. doi: 10.1007/s11239-011-0657-7. PMID 22094974